CLINICAL TRIAL: NCT02119260
Title: A Sponsor Un-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Repeat, Ascending Doses of GSK2798745 in Healthy Subjects and Stable Heart Failure Patients
Brief Title: A First Time in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK2798745 in Healthy Subjects and Stable Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 117387
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-06

CONDITIONS: Oedema, Pulmonary
Keywords: First Time in Human; TRPV4 inhibitor; Heart failure
MeSH Terms: conditions — Pulmonary Edema; Heart Failure | interventions — GSK2798745

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Eight subjects will be randomized to 1 of 4 placebo-controlled dose sequences with 2 subjects in each sequence and each subject having four dose periods (3 active dose of GSK2798745 + 1 placebo dose). GSK2798745 will be administered in a liquid form (suspension or solution) in this cohort. In each treatment period, the subjects will be fasting from the prior midnight to four hours post-dose (Day 1).
  Interventions: Drug: GSK2798745 solution; Drug: GSK2798745 suspension; Drug: Placebo solution; Drug: Placebo suspension
- Cohort 2 (Experimental): Twelve subjects will receive GSK2798745 in three single-dose treatment periods in a fixed sequence. The actual dose-selected will be determined based on review of emerging safety and exposure data from Cohort 1. The dosing will be done in 3 study periods for investigating bioavailability and food effects. In Period 1, subjects will be fasting from midnight to four hours post-dose and will receive GSK2798745 in a liquid form (suspension or solution). In Period 2, subjects will be fasting from midnight to four hours post-dose and will receive a capsule formulation of GSK2798745. In Period 3, subjects will receive GSK2798745 capsule following a standard high fat/high calorie meal.
  Interventions: Drug: GSK2798745 solution; Drug: GSK2798745 suspension; Drug: GSK2798745 capsule
- Cohort 3 (Experimental): Sixteen subjects will be randomized to 2 repeat dose cohorts with 8 subjects in each cohort in a ratio of 6:2 (treatments: placebo). Food intake timing will be determined based on data from Cohorts 1 and 2 (if Cohort 2 is conducted before Cohort 3). Doses will be administered once daily from Day 1 through Day14. Based on data from Cohort 1, the second dose in the repeat-dose period may be skipped to estimate the time invariance in PK. Dosing may be altered to twice daily based on the results obtained in the initial study cohort. Subjects will be fasted from midnight to 4 hours after dosing on Day 1 and Day 14 that entail serial PK sampling. Meal timings on other days will be based on previous cohort data.
  Interventions: Drug: GSK2798745 solution; Drug: GSK2798745 suspension; Drug: GSK2798745 capsule; Drug: Placebo solution; Drug: Placebo suspension; Drug: Placebo capsule
- Cohort 4 (Experimental): Eighteen stable HF subjects will be randomized in this cohort with a treatment:placebo ratio of 1:1. If required, an additional number of subjects (up to 24 total) will be randomized. An additional separate dose group of approximately 18 to 24 subjects may be randomized to GSK2798745 or placebo to gain additional safety, tolerability,pharmacokinetic and pharmacodynamic information, if needed. The subjects will receive GSK2798745 in a single dose (at least the first 6 subjects) followed by a 7 -days repeat dose. Based on data from the cohorts 1, 2 and 3, the dose will be 2.4 mg (initial) in the first group utilizing the capsule formulation administered with or without food.
  Interventions: Drug: GSK2798745 capsule; Drug: Placebo capsule
- Cohort 5 (Experimental): Eight HF subjects will be randomized in this cohort with a treatment: placebo ratio of 3:1. This cohort will evaluate safety, pharmacokinetics, and lung permeability (DLco and DLno) in a boarder, more general population of patients with HF, NYHA Class II or III. Subjects will receive GSK2798745 or placebo (based on randomization) for 7 days. The dose will be 2.4 mg utilizing the capsule formulation administered with or without food. Subjects will remain in house from Day -1 until Day 4 and be fitted with a remote monitoring device; Day 5, 6 and 8 visits will be in home (on Days 5 and 6, they will receive study medication, collect samples for pharmacokinetic analysis, and assess vital signs); and subjects will return to the clinic for Day 7 visit.
  Interventions: Drug: GSK2798745 capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: GSK2798745 solution — Clear, colourless GSK2798745 (0.1 to 0.4mg) solution in aqueous citrate buffer with 4% captisol
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: GSK2798745 suspension — Aqueous suspension of GSK2798745 (>=0.5 mg)
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: GSK2798745 capsule — White Opaque granule filled capsules of GSK2798745 (>=0.5 mg)
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: Placebo solution — Clear, colourless solution of aqueous citrate buffer with 4% captisol
  Arms: Cohort 1; Cohort 3
Drug: Placebo suspension — Visually matching aqueous suspension of hypromellose acetate succinate powder
  Arms: Cohort 1; Cohort 3
Drug: Placebo capsule — Matching white opaque placebo blend filled capsule
  Arms: Cohort 3; Cohort 4; Cohort 5

SUMMARY:
This study is the first administration of GSK2798745 in humans. This will be a sponsor un-blinded, placebo-controlled study to investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GSK2798745, given as single and repeat oral doses to healthy subjects and stable heart failure (HF) subjects. Approximately 28 healthy subjects will be enrolled in the study cohorts (Cohort 1-3) involving single and repeat dose escalations of GSK2798745, while up to 24 stable heart failure subjects will be enrolled in Cohort 4 involving single and repeat dose administration of GSK2798745, with the dose selected based on data from healthy subject cohorts. This would be followed by enrollment of up to 8 subjects with heart failure in Cohort 5 involving repeat dose administration of GSK2798745. The study duration, including screening and follow-up, is not expected to exceed 17 weeks for subjects in the study (in any cohort).

ELIGIBILITY:
Inclusion Criteria:

For Healthy Subject Cohorts (1-3):

* Male or female 18-75 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on an evaluation including medical history, physical examination, laboratory tests and cardiac evaluation including ECG and echocardiogram. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and Body Mass Index (BMI) within the range 18-32 kilogram/ square meter (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the Investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-International Units per milliliter (mIU/mL) and estradiol <40 picogram/millilitre (pg/mL) [<147 picomoles/liter (pmol/L)] is confirmatory.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 2 weeks post last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on averaged QTc values of triplicate ECGs obtained over a brief recording period: QTc <450 milliseconds (msec); or QTc <480 msec in subjects with Bundle Branch Block.

For Heart Failure Subjects (Cohorts 4 and 5):

* Established diagnosis of mild or moderate heart failure of any aetiology with symptoms defined as corresponding to the New York Heart Association (NYHA) Class II or III on stable heart failure therapy for at least 1 month and was not hospitalized for HF for the last three months.
* Male or female 18 years or older, age inclusive, at the time of signing the informed consent.
* ALT, alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on averaged QTc values of triplicate ECGs obtained over a brief recording period: QTc <450msec; or QTc <480msec in subjects with Bundle Branch Block.
* Female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the Investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40mIU/mL and estradiol <40pg/mL (<147pmol/L) is confirmatory.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 2 weeks post-last dose.
* Body weight >=50kg and BMI within the range 18-40kg/m^2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 6 months.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240mL) of beer, 1 glass (125mL) of wine or 1 (25mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator and/or GSK Medical Monitor, contraindicates their participation.
* History of seizure disorder and or stroke within the last 5 years.
* Active ulcer disease or gastrointestinal (GI) bleeding.
* Current smokers (Cohorts 1-4 only).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* A screening cardiac Troponin (cTn) level >ULN.
* Baseline presence of severe aortic stenosis.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Left ventricular ejection fraction <50 percent - (Healthy subjects only).
* Subject who, in the Investigator/designee's judgement, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any evidence of suicidal ideation on any questionnaires e.g., Type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the last 5 years.

For Heart Failure Subjects (Cohort 4):

* History of known primary pulmonary disease requiring current medication or other therapy.
* Orthopnoea of sufficient severity to preclude supine scanning as determined at screening.
* Uncontrolled hypertension (resting systolic blood pressure [BP] > 160 millimeters of mercury [mmHg] or resting diastolic BP > 100 mmHg).
* Resting hypoxia while breathing room air (Peripheral capillary oxygen saturation [SpO2] <88 percent).
* Estimated creatinine clearance (Cockcroft-Gault) <40 mL/minute.
* Contraindication to magnetic resonance imaging (MRI) contrast agents.
* Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes but is not limited to: a. Intracranial aneurysm clips (except Sugita^®; trademark owned by Mizuho Ikakogyo Co.Ltd. Tokyo) or other metallic objects; b. Intra- orbital metal fragments that have not been removed; c. Pacemakers or other implanted cardiac rhythm management/monitoring devices and non-MR conditional heart valves; d. Inner ear implants; and e. History of claustrophobia.

For Heart Failure Subjects (Cohort 5):

* Uncontrolled hypertension (resting SBP >160 mmHg or reporting DBP >100 mmHg).
* Resting hypoxia while breathing room air (SpO2 <88 percent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2016-12-25 (Actual); Study Completion 2016-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Goyal N, Skrdla P, Schroyer R, Kumar S, Fernando D, Oughton A, Norton N, Sprecher DL, Cheriyan J. Clinical Pharmacokinetics, Safety, and Tolerability of a Novel, First-in-Class TRPV4 Ion Channel Inhibitor, GSK2798745, in Healthy and Heart Failure Subjects. Am J Cardiovasc Drugs. 2019 Jun;19(3):335-342. doi: 10.1007/s40256-018-00320-6. PMID 30637626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single dose (SD) and repeat, ascending doses (RD) of GSK2798745 in healthy participants (par.) and stable heart failure par. This study was conducted at two centers in the United Kingdom
Pre-assignment Details: Sixty one par. entered this 5-cohort study where Cohorts 1-3 were healthy par. and Cohorts 4 and 5 were par. with stable heart failure. Of those,1 par. was withdrawn pre-dose due to issues with ECG values. In Cohort 1 and 2, par. were randomized to sequence and in Cohorts 3, 4 and 5 par. were randomized to drug or placebo
Groups:
- Cohort 1: Healthy participants received single oral doses of GSK2798745 0.25 milligram (mg), 1 mg, 5 mg, 12.5 mg and one dose of GSK2798745 matching placebo in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid form (suspension) in this single dose escalation cohort.
- Cohort 2: Healthy participants received three single oral doses of GSK2798745 5 mg in fasted state and following a standard meal. GSK2798745 was administered in a liquid suspension and capsule formulation to evaluate food effect and relative bioavailability.
- Cohort 3: Healthy participants received repeat oral doses of GSK2798745 5 mg or matching placebo (ratio 3:1) in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid formulation (suspension)
- Cohort 4 (GSK2798745 2.4 mg SD and RD): Participants with heart failure received single oral and subsequent 7-days repeat-dose evaluation of GSK2798745 2.4 mg . GSK2798745 was administered in capsule formulation
- Cohort 4 (Placebo RD); Cohort 5 (Placebo RD): Participants with heart failure received placebo. Placebo was administered in capsule formulation
- Cohort 5 (GSK2798745 2.4 mg RD): Participants with heart failure received repeat-doses of GSK2798745 2.4 mg. GSK2798745 was administered in capsule formulation
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 (GSK2798745 2.4 mg SD and RD) | Cohort 4 (Placebo RD) | Cohort 5 (GSK2798745 2.4 mg RD) | Cohort 5 (Placebo RD)
Started | 9 | 12 | 8 | 10 | 13 | 6 | 2
Completed | 8 | 11 | 7 | 10 | 13 | 6 | 2
Not Completed | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 (GSK2798745 2.4 mg SD and RD) | Cohort 4 (Placebo RD) | Cohort 5 (GSK2798745 2.4 mg RD) | Cohort 5 (Placebo RD) | Total
Number analyzed (Participants) | 9 | 12 | 8 | 10 | 13 | 6 | 2 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (6.40) | 42.8 (10.50) | 43.0 (10.43) | 71.0 (7.18) | 64.1 (7.87) | 70.7 (6.92) | 54.0 (9.90) | 55.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 7
  Male | 9 | 12 | 8 | 8 | 8 | 6 | 2 | 53
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian - Central/South Asian Heritage | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White-White/Caucasian/European Heritage | 8 | 12 | 6 | 10 | 11 | 6 | 2 | 55
  African American/African Heritage & White | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Asian & White | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vital Sign Values of Potential Clinical Concern in Healthy Participants
Description: Vital signs included seated supine systolic blood pressure (SBP) and diastolic blood pressure (DBP), heart rate (HR), and respiratory rate (RR). Vital signs criteria of potential clinical concern were SBP: <100 and >170 millimeters of mercury (mmHg); DBP: <50 and >110 mmHg and HR: <50 and >120 beats per minute (bpm). Only those parameters for which at least one value of potential clinical concern was reported are summarized. All Subjects Population includes any participant enrolled into the study who received at least one dose of study medication within a cohort
Time Frame: Up to 17 Weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants
  SBP | 0 | 0 | 8
  DBP | 0 | 0 | 3
  HR | 0 | 0 | 8

2. Primary Outcome: Number of Participants With Vital Sign Values of Potential Clinical Concern in Stable Heart Failure Participants
Description: as for outcome 1
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 4 (GSK2798745 2.4 mg SD and RD) | Cohort 4 (Placebo RD) | Cohort 5 (GSK2798745 2.4 mg RD) | Cohort 5 (Placebo RD)
Number analyzed (Participants) | 10 | 13 | 6 | 2
Participants
  SBP | 7 | 6 | 4 | 1
  DBP | 2 | 0 | 1 | 0
  HR | 4 | 5 | 0 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern in Healthy Participants
Description: ECGs will be obtained in the semi-supine position after at least 5 minutes. The potential clinical concern range for ECG parameters are: QRS interval: >200 milliseconds (msec); time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Bazett's formula (QTcB):>500msec; time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTcF interval): >500 msec; PR interval:>300msec. The number of participants with ECG values of potential clinical concern have been presented.
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants | 4 | 7 | 2

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern in Stable Heart Failure Participants
Description: as for outcome 3
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Groups:
- Cohort 4: Participants with heart failure received single oral and subsequent 7-days repeat-dose evaluation of GSK2798745 2.4 mg or placebo in capsule formulation
- Cohort 5: Participants with heart failure received repeat-doses of GSK2798745 2.4 mg or placebo in capsule formulation
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 23 | 8
Participants | 10 | 3

5. Primary Outcome: Number of Participants With Clinical Chemistry Laboratory Values of Potential Clinical Concern in Healthy Participants
Description: Blood samples were collected from participants to evaluate clinical parameters of potential clinical concern. Clinical parameters included blood urea nitrogen, potassium, total and direct bilirubin, creatinine chloride, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase, alkaline phosphatase, uric acid, glucose, fasting troponin, albumin, sodium calcium total protein, and creatine phosphokinase. The number of participants with clinical chemistry values of potential clinical concern have been presented.
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants | 3 | 6 | 4

6. Primary Outcome: Number of Participants With Clinical Chemistry Laboratory Values of Potential Clinical Concern in Stable Heart Failure Participants
Description: as for outcome 5
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 23 | 8
Participants | 4 | 3

7. Primary Outcome: Number of Participants With Hematology Parameter Laboratory Values of Potential Clinical Concern in Healthy Participants
Description: Blood samples were collected from participants to evaluate hematology parameters of potential clinical concern. Hematology parameters included platelet count, red blood cells count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, neutrophils, white blood cells count, lymphocytes, reticulocyte count, monocytes, hemoglobin, eosinophil, hematocrit, and basophiles. The number of participants with hematology values of potential clinical concern have been presented.
Time Frame: Up to 17 weeks
Population: All subjects population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants | 1 | 3 | 1

8. Primary Outcome: Number of Participants With Hematology Parameter Laboratory Values of Potential Clinical Concern in Stable Heart Failure Participants
Description: as for outcome 7
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 23 | 8
Participants | 3 | 1

9. Primary Outcome: Number of Participants With Abnormal Routine Urinalysis in Healthy Participants
Description: Urine samples were collected to analyze specific gravity, determining potential of hydrogen (pH), glucose, protein, blood, and ketones by dipstick method, and microscopic examination (if blood or protein is abnormal). The number of participants with abnormal urinalysis data have been presented.
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants | 4 | 3 | 2

10. Primary Outcome: Number of Participants With Abnormal Routine Urinalysis in Stable Heart Failure Participants
Description: as for outcome 9
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 23 | 8
Participants | 14 | 3

11. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) in Healthy Participants
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect, any other situation according to medical or scientific judgment, or is associated with liver injury and impaired liver function will be categorized as SAE.
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 9 | 12 | 8
Participants
  Any AE | 5 | 7 | 6
  Any SAE | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) in Stable Heart Failure Participants
Description: as for outcome 11
Time Frame: Up to 17 weeks
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 23 | 8
Participants
  Any AE | 22 | 8
  Any SAE | 0 | 0

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (AUC[0-inf]) Following Single and Repeat Doses of GSK2798745 in Healthy Subjects
Description: Blood samples for Pharmacokinetic (PK) analysis were obtained at Day 1 of each treatment period for analysis of AUC[0-inf]. Log untransformed values for AUC[0-inf] has been presented. The 'PK Population' includes 'All Subjects' population for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Day 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Co 1 (GSK2798745 0.25 mg): Healthy participants received single oral doses of GSK2798745 0.25 mg and one dose of GSK2798745 matching placebo in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid form (suspension) in this single dose escalation cohort.
- Co 1 (GSK2798745 1 mg): Healthy participants received single oral doses of GSK2798745 1 mg and one dose of GSK2798745 matching placebo in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid form (suspension) in this single dose escalation cohort.
- Co 1 (GSK2798745 5 mg): Healthy participants received single oral doses of GSK2798745 5 mg and one dose of GSK2798745 matching placebo in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid form (suspension) in this single dose escalation cohort.
- Co 1 (GSK2798745 12.5 mg): Healthy participants received single oral doses of GSK2798745 12.5 mg and one dose of GSK2798745 matching placebo in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid form (suspension) in this single dose escalation cohort.
- Co 2 (GSK2798745 Fasted Suspension): Healthy participants received three single oral doses of GSK2798745 5 mg in fasted state. GSK2798745 was administered in a liquid suspension to evaluate food effect and relative bioavailability.
- Co 2 (GSK2798745 Fasted Capsule): Healthy participants received three single oral doses of GSK2798745 5 mg in fasted state. GSK2798745 was administered in a capsule formulation to evaluate food effect and relative bioavailability.
- Co 2 (GSK2798745 Fed Capsule): Healthy participants received three single oral doses of GSK2798745 5 mg following a standard meal. GSK2798745 was administered in a capsule formulation to evaluate food effect and relative bioavailability.
- Co 3 (GSK2798745 Day 1-5mg): Healthy participants received oral doses of GSK2798745 5 mg or matching placebo (ratio 3:1) in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid formulation (suspension)
- Co 3 (GSK2798745 Day 14-5mg): Healthy participants received repeat oral doses of GSK2798745 5 mg or matching placebo (ratio 3:1) in fasted state. Participants fasted from midnight to four hours post-dose. GSK2798745 was administered in a liquid formulation (suspension)
Arm/Group | Co 1 (GSK2798745 0.25 mg) | Co 1 (GSK2798745 1 mg) | Co 1 (GSK2798745 5 mg) | Co 1 (GSK2798745 12.5 mg) | Co 2 (GSK2798745 Fasted Suspension) | Co 2 (GSK2798745 Fasted Capsule) | Co 2 (GSK2798745 Fed Capsule) | Co 3 (GSK2798745 Day 1-5mg) | Co 3 (GSK2798745 Day 14-5mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 11 | 11 | 6 | 3
hour*nanogram per milliliter (h*ng/mL) | 9.6 (3.7) | 62.2 (26.6) | 347.0 (122.8) | 686.1 (275.0) | 287.7 (101.2) | 312.1 (71.0) | 361.8 (99.4) | 223.2 (31.0) | 318.7 (39.6)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single and Repeat Dose Administration of GSK2798745 in Healthy Participants
Description: Blood samples for PK analysis were obtained at Day 1 and Day 14 of each treatment period for analysis of Cmax. Log transformed values for Cmax has been presented.
Time Frame: Day 1 (Cohort 1,2,3) and Day 14 (Cohort 3)
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Co 1 (GSK2798745 0.25 mg) | Co 1 (GSK2798745 1 mg) | Co 1 (GSK2798745 5 mg) | Co 1 (GSK2798745 12.5 mg) | Co 2 (GSK2798745 Fasted Suspension) | Co 2 (GSK2798745 Fasted Capsule) | Co 2 (GSK2798745 Fed Capsule) | Co 3 (GSK2798745 Day 1-5mg) | Co 3 (GSK2798745 Day 14-5mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 11 | 11 | 6 | 3
ng/mL | 1.1 (0.4) | 4.2 (1.9) | 22.9 (2.4) | 47.9 (12.1) | 22.2 (5.7) | 23.1 (4.3) | 25.7 (7.9) | 23.9 (5.6) | 29.9 (3.9)

15. Secondary Outcome: Time to Occurrence of Cmax (Tmax) Following Single and Repeat Doses of GSK2798745 in Healthy Participants
Description: Blood samples for PK analysis were obtained at Day 1 of each treatment period and Day 14 of Cohort 3 for analysis of tmax. Log untransformed values for tmax has been presented.
Time Frame: Day 1 (Cohort 1,2,3) and Day 14 (Cohort 3)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: hours
Arm/Group | Co 1 (GSK2798745 0.25 mg) | Co 1 (GSK2798745 1 mg) | Co 1 (GSK2798745 5 mg) | Co 1 (GSK2798745 12.5 mg) | Co 2 (GSK2798745 Fasted Suspension) | Co 2 (GSK2798745 Fasted Capsule) | Co 2 (GSK2798745 Fed Capsule) | Co 3 (GSK2798745 Day 1-5mg) | Co 3 (GSK2798745 Day 14-5mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 11 | 11 | 6 | 3
hours | 1.3 [1 to 2] | 1.6 [1 to 3] | 2.3 [2 to 3] | 2.5 [2 to 3] | 2.0 [1 to 3] | 1.5 [1 to 4] | 1.5 [1 to 3] | 1.8 [1.8 to 3] | 2.0 [2 to 2]

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single and Repeat Dose Administration of GSK2798745 in Stable Heart Failure Participants
Description: Blood samples for PK analysis were obtained at Day 1 and Day 7 of each treatment period for analysis of Cmax. Log untransformed values for Cmax has been presented.
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 8
ng/mL
  Day 1 | 13.7 (1.9) | 13.4 (4.1)
  Day 7 | 17.1 (7.3) | 16.2 (3.5)

17. Secondary Outcome: Area Under the Concentration-time Curve From Pre-dose to 24 Hours Post-dose (AUC [0-24]) Following Single and Repeat Doses of GSK2798745 in Stable Heart Failure Participants
Description: Blood samples for PK analysis were obtained at Day 1 and Day 7 of each treatment period for analysis of AUC (0-24). Log untransformed values for Cmax has been presented.
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 8
hour*ng/mL
  Day 1 | 133.6 (57.9) | 131.4 (11.5)
  Day 7 | 208.5 (115.2) | 207.6 (36.6)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the Follow up (Up to 17 weeks)
Description: AEs and SAEs were collected in All Subjects Population which comprised all the participants enrolled into the study and received at least one dose of study medication within a cohort
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/8 | 0/23 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/8 | 0/23 | 0/8
Other Adverse Events (participants affected / at risk) | 5/9 | 7/12 | 6/8 | 22/23 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=9) | Cohort 2 (N=12) | Cohort 3 (N=8) | Cohort 4 (N=23) | Cohort 5 (N=8)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 2 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (18) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Audiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.